CLINICAL TRIAL: NCT06058871
Title: Ecological Momentary Breastfeeding Intervention to Improve Breastfeeding Outcomes: a Randomized Controlled Trial
Brief Title: Ecological Momentary Breastfeeding Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EMB-RCT1
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-09

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMI intervention group (Experimental): Participants in the intervention group will receive instant messaging (i.e., an EMI delivery platform). Our multidisciplinary team, including an obstetrician, midwife, lactation consultant, biostatistician, and social psychologist, will develop a message library and protocol for EMI delivery.
  Interventions: Behavioral: Regular messages; Behavioral: Nurse-led real-time support messages (chat type)
- Control group (No Intervention): Participants in the control group will receive text messages containing general information on breastfeeding from the Hospital Authority, which is open to the public and includes reminder text messages of important follow-up surveys. Messages will not be personalised, and nurse-led real-time support messages will not be available.

INTERVENTIONS:
Behavioral: Regular messages — The EMI-I messages will be delivered in sequence over three months. The content, frequency, and timing of the messages will be determined by participant preferences, as determined during the baseline evaluation, as personalisation is central to such cognitive and behavioural changes. The messages will mainly be text-based, but other forms such as videos will also be used, depending on the needs of the participants.
  Arms: EMI intervention group
Behavioral: Nurse-led real-time support messages (chat type) — The nurse will initiate 10-15-minute chats via an online platform (e.g., WhatsApp) after all instant messages for each session have been delivered. The nurse will guide the participants to set goals for breastfeeding. Any anticipated barriers will be discussed. The participants can also initiate the chats. While there is no limit to the number of chat messages, nurse-led real-time support messages will be provided during working hours (i.e., 9 am-6 pm on weekdays).
  Arms: EMI intervention group

SUMMARY:
During Chinese mothers' doing the month, they are often housebound and find it difficult to attend group support or seek help during the first month postpartum which is the critical period in sustaining exclusive breastfeeding and at high risk of weaning. This can adversely affect their general well-being, and are associated with stress, anxiety and postnatal depression. Thus, mothers have expressed the need for real-time, real world, personalized support that allow them to get immediate breastfeeding support, helps in overcoming the challenges and subsequently improve exclusive breastfeeding. The aim of the proposed study is to assess the effectiveness of an ecological momentary intervention (EMI)-based breastfeeding intervention in improving exclusive breastfeeding outcomes and to inform clinical practice and services for breastfeeding mothers in Hong Kong. Such interventions have been considered as a rising shift from traditional model of care towards an e-technology based health model that may improve exclusive breastfeeding duration globally.

DETAILED DESCRIPTION:
It is well recognised that breastfeeding is extremely beneficial for child survival, growth, and maternal health and is one of the most effective health interventions for preventing infant and child mortality and promoting lifelong maternal health. In addition, breastfeeding provides significant economic benefits and improves health equity in society. In Hong Kong, data from 2021 shows only 22% of women exclusively breastfeed until six months postpartum, significantly less than both the average global rate of 38% and the World Health Organization (WHO) 2025 target of 50%. Some of the common reasons cited by mothers for early weaning relate to breastfeeding problems that are easily avoided with appropriate early professional support, such as perceived insufficient milk, poor latching and sore breasts. Timely breastfeeding support could therefore promote exclusive breastfeeding. However, such support is often inadequate and has been difficult to obtain during the recent COVID-19 pandemic. In addition, mothers in Hong Kong may find it difficult to leave home during the early postpartum period due to the overwhelming workload and the cultural tradition practice of 'doing the month' in which women remain housebound during the first month postpartum. Therefore, it is be important to provide adequate support to mothers in Hong Kong to ensure that breastfeeding can continue for the optimal duration, thereby providing life-long protection for both mother and infant.

Social cognitive theory (SCT) is widely used to analyse behavioural changes in breastfeeding in response to technology-guided interventions. We will use SCT as a theoretical framework to guide the development of a message library and the delivery of both regular and chat-style support messages. The increased accessibility of an Internet-delivered intervention provides a way to promote each mother's sense of agency by enabling them to access the support they require when they need it. As more people turn to eHealth, the development of an Internet-delivered SCT-based intervention (iSCT-I) to support and educate women may provide a cost-effective way to increase breastfeeding rates. Moreover, the WHO has concluded that will not be possible to reach universal health care coverage without investing in, and broadly adopting, eHealth. EMI is a cost-effective intervention framework that allows personalisation of both the content and delivery method, it can therefore provide a practical and effective strategy for delivering iSCT-I for improving breastfeeding duration and uptake. However, there have been no previous studies of EMI-based breastfeeding interventions. Therefore, we propose an RCT to evaluate the effectiveness of EMI-delivered iSCT-I; a real-time, personalized, and cost-effective approach for improving exclusive breastfeeding rates.

This multi-center randomized control trial adopts two arm design to examine and compare the effects between ecological momentary intervention and usual care to improve breastfeeding outcomes. The study hypotheses are (1) Primiparous mothers who receive an EMI-based breastfeeding intervention will significantly increase their exclusive breastfeeding intention and duration, and (2) The intervention group will have a higher breastfeeding self-efficacy score (BSES) and breastfeeding knowledge and attitude scores at three months postpartum.

A pilot study will be conducted. Aiming to recruit 20 participants. (10:Intervention; 10 Control)

ELIGIBILITY:
Inclusion Criteria:

* be primiparous mothers
* have had a singleton pregnancy and live birth
* have birthed a full-term infant (37-42 weeks gestation)
* speak Cantonese
* be a Hong Kong resident
* have no serious medical or obstetrical complications and have not had their infant admitted to the neonatal intensive care unit (NICU)

Exclusion Criteria:

* is < 37 weeks gestation
* has an Apgar score < 8 at five minutes
* has a birthweight < 2500 grams
* is born with any severe medical conditions or congenital malformations
* is placed in the special care nursery for more than 48 hours after delivery
* is placed in the intensive care nursery after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants in each study groups exclusively breastfeeding | At 1, 2, 3 and 6 months postpartum
  The number of participants who are exclusively breastfeeding at each time point.
Overall duration of any breastfeeding in each study groups | At 1, 2, 3 and 6 months postpartum
  The number of participants who are any breastfeeding at each time point.

SECONDARY OUTCOMES:
Breastfeeding self-efficacy scores between the two study groups | baseline and 1 and 3 months postpartum
  Breastfeeding efficacy measured using Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF). BSES-SF is a 14-item scale with total score ranging from 14 to 70. A higher score indicates higher breastfeeding self-efficacy.
Infant feeding knowledge and attitude scores between the two study groups | baseline and 1 and 3 months postpartum
  Attitude towards breastfeeding measured using the Iowa Infant Feeding Attitude Scale (IIFAS). IIFAS is a 17-item scale with total score ranging from 17 to 85. A higher score indicates a more favorable attitude towards breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Kris YW Dr Lok, PhD, Principal Investigator — School of Nursing, HKU
Locations (2):
- Hong Kong (2):
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No